CLINICAL TRIAL: NCT04178876
Title: Comparison of Laparoscopic Endometrioma Stripping Versus Ethanol Sclerotherapy: Impact on Ovarian Reserve.
Brief Title: Comparison of Laparoscopic Endometrioma Stripping Versus Ethanol Sclerotherapy( CLESS)
Acronym: CLESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2690
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Endometrioma
Keywords: endometrioma; ethanol; sclerotherapy; aspiration; ovarian reserve; endometriosis; AMH
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspiration and Sclerotherapy of endometriomas (Experimental): Aspiration and Sclerotherapy During Laparoscopy Using 95% Ethanol for the Treatment of Endometriomas
  Interventions: Procedure: ethanol sclerotherapy
- laparoscopic stripping technique (Active Comparator): cystectomy of endometriomas during laparoscopy
  Interventions: Procedure: stripping technique

INTERVENTIONS:
Procedure: ethanol sclerotherapy — Endometrioma laparoscopic aspiration and sclerotherapy using 95% ethanol
  Arms: Aspiration and Sclerotherapy of endometriomas
Procedure: stripping technique — Endometrioma laparoscopic cystectomy
  Arms: laparoscopic stripping technique

SUMMARY:
The aim of this study is to compare two different laparoscopic surgical techniques (endometrioma stripping vs ethanol sclerotherapy) in terms of ovarian reserve (AMH levels), recurrence rate and pain relief.

DETAILED DESCRIPTION:
Patients with pelvic pain (VAS score≥4) and ultrasound diagnosis of endometrioma > 4cm candidate to surgical removal of endometrioma will be randomized into 2 group. One Group will undergo laparoscopical stripping technique; the other one will undergo laparoscopic aspiration and sclerotherapy using 95% ethanol.

The women will be introduced with both operative options and they will be informed about the randomization . After an elaborate explanation about the study they will sign an informed consent form. the following data will be collected prior the operation: age, gravity & parity, operative history, general medical history, the cyst size, AMH (Anti Mullerian Hormone), symptoms related to endometriosis (through VAS score), fertility history including any fertility treatment in the past and planned pregnancy after the operation.

The laparoscopy will take place in Fondazione Policlinico Gemelli IRCSS, Roma. in the study group the cyst content will be aspirated and flushed with normal saline. 95% sterile ethanol will be instilled into the cyst through a Nelathon catheter. Ethanol will be left in the cyst for 15 min then aspirated as completely as possible following normal saline flushing. In the control group we will follow the standard treatment which is cystectomy.

The women will be followed at 1 , 3 , 6 and 12 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18-35 years old
* Women with ultrasound diagnosis of ovarian endometrioma ≥4cm (with or without deep infiltrating endometriosis)
* History of dysmenorrhea and/or chronic pelvic pain
* candidates for elective laparoscopy due to endometriosis.

Exclusion Criteria:

* - Previous surgery for ovarian endometriosis
* Evidence of premature ovarian failure (follicle stimulating hormone ≥40 international units/L)
* Endocrinal disorders that might affect ovarian function (e.g., polycystic ovary syndrome, thyroid dysfunction, hyperprolactinemia)
* Ultrasound suspicious of ovarian malignant disease according IOTA criteria
* endometrial cyst < 4 cm. • ethanol sensitivity.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This is a Gynecological study
Enrollment: 64 (Estimated)
Dates: Start 2019-09-13 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
impact on ovarian reserve, in terms of reduction of serum AMH levels | up to 12 months after the laparoscopy
  The AMH levels will be evaluated 1 month before the surgery and 1, 6 and 12 months after surgery.

SECONDARY OUTCOMES:
endometrioma recurrence rate for the two surgical techniques | up to 12 months after the laparoscopy
  Ultrasound examination that demonstrate the presence/lack of ovarian cyst with sonographic features of endometrioma in the ovary where the procedure took place.
pain relief after surgery | up to 12 months after the laparoscopy
  The severity of pelvic pain , assessed using a visual analogue scale with no-pain classified as 0 and worst imaginable pain as 10.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, MD, Principal Investigator — Fondazione Policlinico Gemelli, IRCSS Università Cattolica del Sacro Cuore, Roma
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: data will become available following publication.
Access Criteria: To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Sweed MS, Makled AK, El-Sayed MA, Shawky ME, Abd-Elhady HA, Mansour AM, Mohamed RM, Hemeda H, Nasr-Eldin EA, Attia NS, Eltaieb E, Allam H, Hussein A. Ovarian Reserve Following Laparoscopic Ovarian Cystectomy vs Cyst Deroofing for Endometriomas. J Minim Invasive Gynecol. 2019 Jul-Aug;26(5):877-882. doi: 10.1016/j.jmig.2018.06.022. Epub 2018 Sep 5. PMID 30193971
- [Background] Cohen A, Almog B, Tulandi T. Sclerotherapy in the management of ovarian endometrioma: systematic review and meta-analysis. Fertil Steril. 2017 Jul;108(1):117-124.e5. doi: 10.1016/j.fertnstert.2017.05.015. Epub 2017 Jun 1. PMID 28579409
- [Background] Messalli EM, Cobellis G, Pecori E, Pierno G, Scaffa C, Stradella L, Cobellis L. Alcohol sclerosis of endometriomas after ultrasound-guided aspiration. Minerva Ginecol. 2003 Aug;55(4):359-62. PMID 14581861
- [Background] Garcia-Tejedor A, Castellarnau M, Ponce J, Fernandez ME, Burdio F. Ethanol sclerotherapy of ovarian endometrioma: a safe and effective minimal invasive procedure. Preliminary results. Eur J Obstet Gynecol Reprod Biol. 2015 Apr;187:25-9. doi: 10.1016/j.ejogrb.2015.02.004. Epub 2015 Feb 16. PMID 25739052
- [Background] Kovacevic VM, Andelic LM, Mitrovic Jovanovic A. Changes in serum antimullerian hormone levels in patients 6 and 12 months after endometrioma stripping surgery. Fertil Steril. 2018 Nov;110(6):1173-1180. doi: 10.1016/j.fertnstert.2018.07.019. PMID 30396562